CLINICAL TRIAL: NCT05991271
Title: Multicenter Pivotal Study to Evaluate the Treatment of Severe Aortic Valve Stenosis With Next-Generation Venus-Vitae Transcatheter Heart Valve (THV) System
Brief Title: Venus-Vitae Pivotal Study Smart-Align Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Venus MedTech (HangZhou) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTAR-23-03
Record Dates: First submitted 2023-06-26; First posted 2023-08-14 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- procedure (Experimental): implant valve by TAVR
  Interventions: Device: Venus-Vitae Transcatheter Heart Valve System

INTERVENTIONS:
Device: Venus-Vitae Transcatheter Heart Valve System — The Venus-Vitae THV is comprised of balloon-expandable and radiopaque cobalt-chromium alloy frame, porcine pericardium tri-leaflet, porcine pericardium inner skirt, polyurethane outer skirt, PTFE assembly sutures, and three radiopaque gold markers (Figure 1). The valve utilizes Venus Endura technology and stored in a non-aqueous condition.

SUMMARY:
The purpose is to evaluate the safety, effectiveness and performance of Venus-Vitae Transcatheter Heart Valve System in patients with severe aortic stenosis.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, non-randomized interventional study to evaluate the safety, effectiveness and performance of the Venus-Vitae Transcatheter Heart Valve System in patients with severe aortic stenosis. Clinical visits will be scheduled at screening, pre-discharge, 30 days, 6 months, 12 months and annually thereafter to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with the symptoms of severe aortic stenosis
3. Severe aortic stenosis (AS, grade 3+), defined as AVA ≤ 1 cm2 (AVAi ≤ 0.6 cm2/m3) or Vmax ≥ 4.0 m/s or MPG ≥ 40 mmHg determined by echocardiography
4. Patients deemed for cardiac intervention by a heart team
5. Patients of all surgical risk categories can be enrolled in this study, but should follows local medical practices and regulatories.
6. Patients or their legal reprensentatives are willing to participate in the study and provide written informed consent, and agree to follow the follow-up requirements

Exclusion Criteria:

A subject meeting any of the following criteria shall be excluded:

Co-morbidities

1. Previous mechanical or biological aortic valve replacement
2. Untreated mitral, tricuspid or pulmonary valve diseases requiring procedural intervention
3. Acute myocardial infact within 30 days prior to index procedure
4. Untreated clinical significant coronary artery disease requiring revascularization
5. Any therapeutic invasive cardiac procedure performed within 30 days (or drug-eluting coronary stent/scaffold implant within 6 months)
6. Sever symptomatic carotid artery stenosis
7. Stroke or TIA within 3 months or Modified Rankin Scale ≥ 4 disability
8. Chronic kidney disease (eGFR<30 mL/min/1.73m2)
9. Haemotologic disorders: Leukopenia (WBC < 3000 cell/mL), anemia (Hgb < 9 g/dL), thrombocytopenia (Plt< 50,000 cell/mL), or any known blood clotting disorder, deemed clinically significant after consultation with Haematooncology specialists
10. Severe right heart dysfunction Anatomical
11. LVEF < 20%
12. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation
13. Inappropriate anatomy for femoral introduction and delivery of study device
14. Native aortic valve geometry and size unfavorable for study device anchoring General
15. Haemodynamics instability requiring inotropic support or intra-aortic balloon pump (IABP) or other hemodynamic support device, or any mechanical heart assistance
16. Known hypersensitivity or contraindication to antiplatelet, antithrombotic medications, or cobalt-chromium leading to be unable to undergo index procedure per physicians' judgement
17. Life expectancy ≤ 1 year due to noncardiac reasons
18. Active infection requiring antibiotic therapy including infective endocarditis
19. Planned relevant concomitant procedure within 30 days post index procedure
20. Pregnant, breastfeeding or intend to become pregnant within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
The rate of deaths at the one-year follow-up visit post procedure | 1 Years
  All-cause mortality (The rate of deaths at the one-year follow-up visit post procedure)
Acceptable Hemodynamic Performance at 30 days | 30 Days
  Acceptable Bio-prosthesis Hemodynamic Performance at 30 days, defined as:
  * Mean gradient < 20mmHg
  * Less than moderate aortic regurgitation (perivalvular and transvalvular)

SECONDARY OUTCOMES:
Occurrence of the following adverse events echocardiogram during follow-up | 5 Years
  Occurrence of the following adverse events echocardiogram during follow-up (The rate of follow events during the follow-up)
  * All-cause mortality
  * All stroke
  * Life-threatening bleeding
  * Acute MI
  * Heart failure hospitalizations
  * New permanent pacemaker implantation
  * Major vascular complication
  * Acute kidney injury
  * Aortic valve re-intervention (surgical or transcatheter)
  * Valve thrombosis
  * Structural valve deterioration
Technical success is defined as the following | During the Procedure
  Technical success (at exit from procedure room) (VARC-3[1]) (The rate of Technical success at the Procedure)
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device or a major vascular or access-related, or cardiac structural complication
The rate of device success is defined as the following | Up to 1 week
  Device success (in-hospital) (VARC-3[1]) (The rate of device success during the in-hospital)
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (mean gradient < 20 mmHg, peak velocity <3 m/s, and less than moderate aortic regurgitation)
The rate of acceptable valve function at pre-discharge by echocardiogram defined as the following: | Up to 1 week
  Acceptable valve function at pre-discharge by echocardiogram (The rate of follow events during the follow-up)
  * Freedom from moderate or greater patient-prosthesis mismatch (PPM)
  * MPG <20mmHg
  * Freedom from moderate or greater regurgitation (transvalvular and paravalvular)
  * Freedom from reoperation or intervention
The rate of freedom from severe coronary overlap assessed by post-implant angiogram | immediately after the procedure
  Freedom from severe coronary overlap assessed by post-implant angiogram
The rate of freedom from mild or greater commissure misalignment assessed by post-implant angiogram and/or 30-day CT | 30-Days
  Freedom from mild or greater commissure misalignment assessed by post-implant angiogram and/or 30-day CT (post-implant 30-day CT scan is not mandatory for each subjects)
The rate of freedom from mild or greater PVL by echocardiogram during follow-up | 5 Years
  Freedom from mild or greater PVL by echocardiogram during follow-up
New York Heart Association (NYHA) classification during follow-up | 5 Years
  New York Heart Association (NYHA) classification during follow-up

IPD SHARING:
Plan to Share IPD: No